CLINICAL TRIAL: NCT06892613
Title: A Comparison of the Effectiveness of Emotion-Focused Couples Therapy and Behavioral Couples Therapy in Reducing Depression and Anxiety Symptoms in Married Couples
Brief Title: EFCT vs. BCT for Depression and Anxiety in Married Couples
Acronym: EFCT-BCT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beykoz University (Other)
Collaborators: Uskudar University (Other); Istanbul Nisantasi University (Other)
Responsible Party: Principal Investigator, Eda Yilmazer, Primary Investigator, Beykoz University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EFCT_BCT_Anxiety_Depression_20
Record Dates: First submitted 2025-02-16; First posted 2025-03-25 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Depression Anxiety Disorder; Anxiety
Keywords: Depression; Anxiety; Emotion-Focused Couples Therapy; Behavioral Couples Therapy; Mental Health; Psychotherapy; Marital Counseling
MeSH Terms: conditions — Anxiety Disorders; Depression; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of three parallel groups: Emotion-Focused Couples Therapy (EFCT), Behavioral Couples Therapy (BCT), or a control group. Each intervention group will receive 12 weekly therapy sessions, while the control group will receive no intervention during the study period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Emotion-Focused Couples Therapy (EFCT) Group (Experimental): Participants in this group will receive Emotion-Focused Couples Therapy, consisting of 12 weekly 50-minute sessions focused on emotional expression, attachment needs, and improving emotional bonds between partners.
  Interventions: Behavioral: Emotion-Focused Couples Therapy (EFCT)
- Behavioral Couples Therapy (BCT) Group (Experimental): Participants in this group will receive Behavioral Couples Therapy, consisting of 12 weekly 50-minute sessions focused on modifying maladaptive behaviors, enhancing communication, and developing problem-solving strategies.
  Interventions: Behavioral: Behavioral Couples Therapy (BCT)
- Control Group (No Intervention): Participants in this group will receive no therapeutic intervention during the study period but will be offered therapy after the study is completed.

INTERVENTIONS:
Behavioral: Emotion-Focused Couples Therapy (EFCT) — EFCT is a structured approach to couples therapy that focuses on helping partners understand and express their emotions, address attachment insecurities, and strengthen their emotional connection.
  Arms: Emotion-Focused Couples Therapy (EFCT) Group
Behavioral: Behavioral Couples Therapy (BCT) — BCT is a form of therapy that aims to improve relationship satisfaction through behavioral change, communication training, and problem-solving techniques.
  Arms: Behavioral Couples Therapy (BCT) Group

SUMMARY:
This study compares the effectiveness of Emotion-Focused Couples Therapy (EFCT) and Behavioral Couples Therapy (BCT) in reducing depression and anxiety symptoms in married couples. A total of 150 married couples aged 18-65 will be screened, and 60 couples with high depression and anxiety levels will be selected. These couples will be randomly assigned to one of three groups: EFCT, BCT, or a control group. Therapy sessions will be conducted weekly for 12 weeks, with assessments before therapy, after the 6th and 12th sessions, and at a 3-month follow-up. The study aims to determine which therapy is more effective in improving mental health outcomes in couples.

DETAILED DESCRIPTION:
Detailed Description:

This randomized controlled trial (RCT) is designed to compare the effectiveness of Emotion-Focused Couples Therapy (EFCT) and Behavioral Couples Therapy (BCT) in reducing depression and anxiety symptoms among married couples. The study will involve 150 married couples aged between 18 and 65, who have been married for at least one year, have no current psychiatric diagnosis, and are not undergoing any form of psychological therapy at the time of recruitment. Recruitment will be conducted through advertisements, social media platforms, and referrals from community centers and family counseling services in Istanbul.

Study Design:

The study will follow a parallel-group design with a 1:1:1 allocation ratio. After an initial screening process, participants will complete a sociodemographic form and two standardized psychological assessments: the Beck Depression Inventory-II (BDI-II) and the Beck Anxiety Inventory (BAI). Based on the assessment results, 60 couples with high levels of depression and anxiety symptoms will be selected for the intervention phase. A computer-generated randomization process will assign 20 couples to the EFCT group, 20 couples to the BCT group, and 20 couples to a control group that will not receive therapy during the study period.

Intervention Protocol:

The EFCT intervention will consist of 12 weekly therapy sessions, each lasting 50 minutes, facilitated by trained clinical psychologists experienced in EFCT. The therapy will focus on enhancing emotional expression, addressing attachment-related insecurities, and fostering emotional bonding between partners. The EFCT framework will follow the standard intervention model, encompassing the three stages of de-escalation, restructuring of interactions, and consolidation.

The BCT intervention will also include 12 weekly 50-minute sessions, focusing on modifying maladaptive behavioral patterns, improving communication, and developing effective problem-solving skills within the relationship. The BCT approach will be guided by the established protocols emphasizing behavioral exchange, communication training, and cognitive restructuring techniques.

The control group will not receive any therapeutic intervention during the 12-week study period but will be offered counseling sessions after the completion of the study to ensure ethical integrity and participant well-being.

Assessment Timeline and Outcome Measures:

Participants will undergo assessments at four key time points:

Baseline (Pre-Intervention): Before the first therapy session, all couples will complete the BDI-II and BAI.

Mid-Intervention: After the 6th therapy session, the BDI-II and BAI will be administered again to evaluate initial changes in depression and anxiety levels.

Post-Intervention: Upon completion of the 12th therapy session, participants will complete the BDI-II and BAI to measure the immediate effects of the intervention.

Follow-Up: Three months after the final therapy session, couples will complete the BDI-II and BAI to assess the sustainability of the therapeutic outcomes.

Data Collection and Management:

Data will be collected using paper-based forms and subsequently entered into a secure electronic database by research assistants. Double data entry will be implemented to minimize errors. All data will be anonymized, and participants will be assigned unique identification codes to ensure confidentiality. The principal investigator will oversee data management and ensure adherence to the study protocol.

Data Analysis Plan:

Statistical analysis will be conducted using SPSS software (version 28.0). Repeated measures ANOVA will be employed to examine within-group and between-group differences over time, focusing on changes in BDI-II and BAI scores. Post-hoc tests (Bonferroni correction) will be used to identify specific differences between the EFCT, BCT, and control groups at each assessment point. Effect sizes (Cohen's d) will be calculated to determine the magnitude of therapeutic effects. Missing data will be handled using multiple imputation methods to maintain the integrity of the dataset.

Ethical Considerations:

The study has received ethical approval from Üsküdar University (Reference number: 61351342/020-675) on December 29, 2024. All participants will provide written informed consent prior to participation. Confidentiality will be maintained throughout the study, and participants will have the right to withdraw at any time without any consequences. The study adheres to the ethical guidelines outlined in the Declaration of Helsinki.

Clinical Significance:

This study aims to provide empirical evidence on the comparative effectiveness of EFCT and BCT in alleviating depression and anxiety symptoms in married couples. The findings are expected to contribute to the development of evidence-based therapeutic interventions in marital counseling, highlighting the potential benefits of both emotion-focused and behavioral approaches in improving mental health and relationship quality.

ELIGIBILITY:
Inclusion Criteria:

* Married couples aged between 18 and 65 years
* Married for at least one year
* No current psychiatric diagnosis or history of psychiatric treatment
* Not receiving any form of psychological therapy at the time of recruitment
* Ability to provide informed consent
* Willingness to participate in all therapy sessions and assessments

Exclusion Criteria:

* Current or past psychiatric diagnosis (excluding mild transient conditions)
* Ongoing psychological therapy or psychiatric treatment
* Severe mental health disorders (e.g., schizophrenia, bipolar disorder), Substance abuse or dependency
* Severe medical conditions that may interfere with participation
* Refusal to participate in follow-up assessments

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-09-15 (Estimated)

PRIMARY OUTCOMES:
The Beck Depression Inventory-II (BDI-II) | Baseline, after the 6th session (6 week), after the 12th session (12 week), and at 3-month follow-up (24 week)
  The Beck Depression Inventory-II (BDI-II) will be used to measure changes in depression symptoms over time. Scores range from 0 to 63, with higher scores indicating more severe depressive symptoms.
The Beck Anxiety Inventory (BAI) | Baseline, after the 6th session (6 week), after the 12th session (12 week), and at 3-month follow-up (24 week)
  The Beck Anxiety Inventory (BAI) will be used to measure changes in anxiety symptoms over time. Scores range from 0 to 63, with higher scores indicating more severe anxiety symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Eda Yılmazer, Phd, Principal Investigator — Beykoz University; Metin Çınaroğlu, Phd, Principal Investigator — Istanbul Nisantasi University; Selami VArol Ülker, Phd, Principal Investigator — Üsküdar University
Locations (1):
- Beykoz University, Istanbul, Istanbul, Turkey (Türkiye)